CLINICAL TRIAL: NCT05048251
Title: Individually Targeted Neuromodulation for Contamination-based Obsessive-compulsive Disorder
Brief Title: Individually Targeted Neuromodulation for Contamination-based OCD
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Mclean Hospital (Other)
Collaborators: Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, Brian P. Brennan, MD, Medical Director, Obsessive-Compulsive Disorder Institute, Mclean Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2021P000141
Record Dates: First submitted 2021-08-27; First posted 2021-09-17 (Actual); Last update posted 2024-03-15 (Actual); Status verified 2024-03

CONDITIONS: Obsessive-Compulsive Disorder
MeSH Terms: conditions — Obsessive-Compulsive Disorder

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (3):
- cTBS (Experimental): continuous TBS to right MFG
  Interventions: Device: cTBS
- iTBS (Experimental): intermittent TBS to right MFG
  Interventions: Device: iTBS
- sham (Sham Comparator): sham stimulation to right MFG
  Interventions: Device: sham

INTERVENTIONS:
Device: cTBS — continuous theta burst stimulation
  Arms: cTBS
Device: iTBS — intermittent theta burst stimulation
  Arms: iTBS
Device: sham — sham stimulation
  Arms: sham

SUMMARY:
Patients with obsessive-compulsive disorder (OCD) experience a wide array of different types of obsessions and compulsions. However, current treatments for OCD employ a "one size fits all" approach and are used for all patients regardless of symptom type. In this project, the investigators propose to investigate whether a novel method of transcranial magnetic stimulation specifically reduces contamination/washing symptoms - one of the most common types of OCD.

DETAILED DESCRIPTION:
The symptoms of obsessive-compulsive disorder (OCD) appear linked to dysfunction in a cortico-striato-thalamo-cortical circuit. However, obsessions and compulsions vary widely among OCD patients, suggesting that other symptom-specific brain networks may accompany this core defect. Identifying such networks could lead to personalized treatments, improving upon current "one size fits all" approaches.

Factor analyses have found distinct symptom dimensions in OCD, but the neural systems specific to these dimensions remain unclear. Using a novel, data-driven, individual-level approach to resting-state functional connectivity magnetic resonance imaging (fcMRI), the investigators have shown that increased connectivity between right medial frontal gyrus (R MFG) and brain regions within the ventral attention network (VAN) - regions critical to reorienting attention in response to relevant external stimuli - specifically predicted the severity of contamination/washing (CONTAM) symptoms, and attenuation of this hyperconnectivity following treatment was associated with improvement in CONTAM symptoms. Based on these findings, the investigators hypothesize that decreasing R MFG-VAN connectivity via transcanial magnetic stimulation (TMS) will normalize attentional reorienting and reduce CONTAM symptoms in individuals with contamination-based OCD.

The investigators propose a two-phase program to investigate R MFG-targeted TMS as a potential intervention for contamination-based OCD. First, in the currently study, the investigators will determine the optimal TMS paradigm to decrease R MFG-VAN connectivity by administering continuous, intermittent, and sham theta burst stimulation (cTBS, iTBS, sham) to individuals with contamination-based OCD using a novel individual-level approach to target the area of R MFG most strongly correlated with VAN based on each participant's pre-treatment connectivity data. Second, the investigators will use the TMS approach identified in this study to test the links between reduced R MFG-VAN connectivity, decreased VAN activation during attentional reorienting, and reduced CONTAM symptoms in a future study using a larger sample of OCD individuals with CONTAM.

ELIGIBILITY:
Inclusion Criteria:

1. male or female age 18-55 years old
2. DSM-5 diagnosis of OCD as primary presenting disorder
3. CONTAM as the predominant symptom dimension (i.e., Dimension 4 (CONTAM symptoms) is the highest score on the Dimensional Yale-Brown Obsessive Compulsive Scale (D-YBOCS); participants with more than one Dimension as highest score will still be eligible as long as Dimension 4 is one of these)
4. score of ≥ 8 on Dimension 4 of the D-YBOCS
5. taking no psychiatric medications or on a stable dose of an SSRI, clomipramine, SNRI, or second generation antipsychotic for at least 4 weeks prior to enrollment. Use of PRN benzodiazepines will be permitted as long as the dose/usage has not changed significantly leading up to enrollment. No medication changes will be permitted during the study
6. have not initiated a new course of exposure and response prevention (ERP) therapy within 4 weeks of enrollment (ongoing ERP will be permitted if initiated more than 8 weeks before enrollment).

Exclusion Criteria:

1. positive urine drug screen (other than prescribed benzodiazepines)
2. use of psychiatric medications other than permitted above
3. substance use disorder in the last 3 months (with the exception of nicotine)
4. history of schizophrenia, bipolar disorder, autism, Tourette's syndrome (current and past history of depressive, anxiety, and eating disorders permitted as long as OCD is considered the primary disorder)
5. active suicidal ideation over the week prior to screening (as indicated by answering yes to questions 1 or 2 on the C-SSRS)
6. history of traumatic brain injury, seizure disorder, neurodegenerative disease, or other organic brain disease
7. pregnancy or lactating
8. contraindication to MRI scanning or TMS

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 50 (Estimated)
Dates: Start 2022-07-01 (Actual); Primary Completion 2024-06-30 (Estimated); Study Completion 2024-06-30 (Estimated)

PRIMARY OUTCOMES:
Functional connectivity between R MFG and brain regions within VAN (expressed as a Z-score) | 6 weeks
  Change in functional connectivity between: 1) R MFG and right temporoparietal junction (R TPJ); 2) R MFG and left temporoparietal junction (L TPJ); 3) R MFG and right inferior frontal gyrus (R IFG); 4) R MFG and left inferior frontal gyrus (L IFG); 5) R MFG and right anterior insula (R AI); 6) R MFG and left anterior insula (L AI); 7) R MFG and right posteromedial putamen; and 8) R MFG and left posteromedial putamen

SECONDARY OUTCOMES:
Functional activation of R MFG and brain regions within VAN during an RSVP task (expressed as a beta value) | 6 weeks
  Change in activation in: 1) R MFG; 2) R TPJ; 3) L TPJ; 4) R IFG; 5) L IFG; 6) R AI; 7) L AI; 8) R posteromedial putamen; and 9) L posteromedial putamen during visual search on the RSVP task
Dimensional Yale-Brown Obsessive Compulsive Scale (D-YBOCS) | 6 weeks
  Change in score on Category 4 (contamination) on the Dimensional Yale-Brown Obsessive Compulsive Scale (D-YBOCS) (minimum score: 0 and maximum score: 18; higher scores represent more severe symptoms)
Yale-Brown Obsessive Compulsive Scale (YBOCS) | 6 weeks
  Change in total score on the Yale-Brown Obsessive Compulsive Scale (YBOCS) (minimum score: 0 and maximum score: 40; higher scores represent more severe symptoms)

CONTACTS AND LOCATIONS:
Overall Officials: Brian P Brennan, MD, Principal Investigator — Mclean Hospital
Locations (1):
- McLean Hospital, Belmont, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No